CLINICAL TRIAL: NCT06191055
Title: Randomized Clinical Trial to Analyze the Efficacy of Chronic Intake of Different Doses of a β-alanine Supplement on Performance in Recreational Cross-country Road Cyclists
Brief Title: Study to Analyze the Efficacy of Chronic Intake With a β-alanine Supplement in Recreational Cyclists
Acronym: B-AC2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Católica San Antonio de Murcia (Other)
Responsible Party: Principal Investigator, Francisco Javier López Román, Principal Investigator, Universidad Católica San Antonio de Murcia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: UCAMCFE-00030
Record Dates: First submitted 2023-12-02; First posted 2024-01-05 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2023-11

CONDITIONS: Beta Alanine Supplementation
Keywords: Chronic effect; Beta Alanine
MeSH Terms: interventions — beta-Alanine; Control Groups

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Beta Alanine high dose (Experimental): Consumption for 28 days.
  Interventions: Dietary Supplement: Beta Alanine high dose
- Beta Alanine low dose (Experimental): Consumption for 28 days.
  Interventions: Dietary Supplement: Beta Alanine low dose
- Control group (Placebo Comparator): Consumption for 28 days.
  Interventions: Other: Control group

INTERVENTIONS:
Dietary Supplement: Beta Alanine high dose — 4 intakes of 5 g of beta alanine every 3 hour.
  Arms: Beta Alanine high dose
Dietary Supplement: Beta Alanine low dose — 4 intakes of 2.5 g of beta alanine every 3 hour.
  Arms: Beta Alanine low dose
Other: Control group — 4 intakes of 2.5 g of wheat semolina every 3 hour.
  Arms: Control group

SUMMARY:
Randomized, controlled, double-blind, single-center, controlled clinical trial with three parallel arms depending on the product consumed (experimental product dose 1 and dose 2 and placebo product) to measure the efficacy of 28-day consumption of a sustained-release beta alanine on the physiological efficacy of physical performance in recreational cyclists.

DETAILED DESCRIPTION:
Subjects meeting the selection criteria will be randomly assigned to each of the study groups (investigational product dose 1 or dose 2, or placebo, depending on the group to which they have been assigned).

The product to be consumed is beta alanine. Participants will consume the product for 28 days. They will have to take 4 intakes every three hours, the first intake being two hours after waking up.

The study subjects will have to make 2 visits to the laboratory. Physical performance and physiological changes will be evaluated with a 10-minute time trial. The first test will be performed without product consumption and the second after 28 days of consumption.

ELIGIBILITY:
Inclusion Criteria:

* Male cyclists with more than two years of cycling experience.
* Perform tests without fatigue.
* Road bike training at least twice a week.

Exclusion Criteria:

* Participants with chronic illness.
* Have a long-term injury that prevents you from training in the previous month.
* Inability to understand informed consent.
* Have consumed beta alanine in the three years prior to the start of the study.
* Consumption of other supplements that may alter performance.

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2023-12-04 (Actual); Primary Completion 2024-02-05 (Actual); Study Completion 2024-03-11 (Actual)

PRIMARY OUTCOMES:
Power | It will be measured on two different occasions. The first day and twenty-eight days later.
  Physical performance is measured by direct variables evaluated by the power roller (average power, maximum power, etc.).
Distance covered | It will be measured on two different occasions. The first day and twenty-eight days later.
  Physical performance is measured by direct variables evaluated by the power roller.

SECONDARY OUTCOMES:
Fatigue | Change of baseline rate of perceived exertion at twenty-eight days
  Rate of perceived exertion
Paresthesia test | It will be measured on two different occasions. on day 1 (before consumption) and twenty-eight days after (after consumption).
  Visual analogue scale (1-10)
Microcapillary blood | It will be measured on two different occasions. Day one and twenty-eight days later.
  This test provides biochemical variables (ABL90FLEX) with 70 ml of capillary blood (Na, K, Glucose, Lactate, etc). It is used to evaluate the effort made by the cyclist.
Lactate | It will be measured on two different occasions. Day one and twenty-eight days later.
  Lactate levels will be measured using the Lactate Pro
Heart Rate | It will be measured on two different occasions. Day one and twenty-eight days later.
  The heart rate will be evaluated by means of a heart rate strap.
Body weight | The test will be measured at baseline and after 28 days of consumption.
  It is a control variable. Measured by bioimpedance.
Fat mass | The test will be measured at baseline and after 28 days of consumption.
  It is a control variable. Measured by bioimpedance.
Muscle mass | The test will be measured at baseline and after 28 days of consumption.
  It is a control variable. Measured by bioimpedance.
Liver safety variables | It will be measured twice, once at baseline or at the end of the study after 28 days.
  It is a blood test that measures the presence of some enzymes, proteins and bilirubin in the blood, with the aim of determining if there is any alteration in the liver. Enzyme GPT, GOT, Gamma GT, LDH, alkaline phosphatase and bilirubin (UI/L)

CONTACTS AND LOCATIONS:
Locations (1):
- Catholic University of Murcia, Murcia, Spain